CLINICAL TRIAL: NCT04388553
Title: Single Shot Lumbar Erector Spinae Plane (ESP) Block in Total Hip Replacement (THR): a Randomized Control Trial
Brief Title: Single Shot Lumbar Erector Spinae Plane (ESP) Block in Total Hip Replacement (THR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Anyon Chan, Principal investigator, Resident Trainee in Department of Anaesthesia and Intensive Care, Tuen Muen Hospital, New Territories West Cluster, HKSAR, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTWC/REC/20007
Record Dates: First submitted 2020-05-09; First posted 2020-05-14 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Total Hip Replacement; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: For the treatment arm, lumbar ESP block is performed while for control arm no regional anaesthesia is performed nor saline is injected into the ESP. Before proceeding to ESP block, the back is cleaned with aseptic technique and draped. 40 mL of 0.25% levobupivacaine (or maximum of 2mg/kg body weight made up to same volume) is injected into the ESP.
Who Masked: Participant, Outcomes Assessor
Masking Description: After the patient is put under GA and turned lateral, the sealed opaque envelope is opened. Unilateral lumbar ESP block is performed in participants under treatment arm, while no regional block is performed for control arm.
  The patient is assessed by an independent assessor from the acute pain service team 24 hours after the operation, who is blinded from the allocation result.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): lumbar ESP block is performed. Before proceeding to ESP block, the back is cleaned with aseptic technique and draped. 40 mL of 0.25% levobupivacaine (or maximum of 2mg/kg body weight made up to same volume) is injected into the ESP.
  Interventions: Procedure: single shot lumbar Erector Spinae Plane block
- Control (No Intervention): no regional anaesthesia is performed nor saline is injected into the ESP

INTERVENTIONS:
Procedure: single shot lumbar Erector Spinae Plane block — unilateral (operative side), performed at L1 level, under ultrasound guidance
  Arms: Treatment

SUMMARY:
Total hip replacement is a common orthopaedic procedure that improves pain and mobility in a variety of pathologies like osteoarthritis, rheumatoid arthritis and avascular necrosis. Post-operative complications, for instance, venous thromboembolism and chest infection have long been documented in literature. These complications can have a bearing on long term survival, and may be prevented by early mobilisation. Therefore, pain control plays an important role in enhancing post-operative recovery, which may also shorten length of stay and reduce overall cost.

Multimodal analgesia is applied to these patient, with combination of opioid, oral adjuvant and regional anaesthesia. Each of the components has its own limitation; for opioid, post-operative nausea and vomiting (PONV) and respiratory depression limits its use, and adjuvants like non-steroidal anti-inflammatory drugs (NSAID) are contraindicated in certain patient populations (renal impairment, ischaemic heart disease, coagulopathy). Various regional techniques like femoral nerve block, fascia iliaca block, lumbar plexus block, paravertebral block and epidural anaesthesia are proposed but may be limited by incomplete coverage (due to the innervation by femoral and obturator nerve for the anterior aspect of the joint and sciatic nerve for the posterior aspect, with contribution of lateral cutaneous nerve of thigh for the wound), the invasive nature of the regional technique (psoas haematoma for lumbar plexus block, epidural haematoma for epidural anaesthesia (EA)) or cardiovascular effects like hypotension from EA.

Erector spinae block, first introduced by in 2016 as a chronic pain intervention, was also used in hip surgery from a case report in 2018. However, currently the evidence for lumbar ESP block is limited mainly to case reports, while randomised control trial is scarce. More concrete data are required to determine the efficacy of this novel technique.

It is postulated that single shot lumbar ESP injected at L1 level can 1) reduced post-operative pain score 2) reduced post-operative 24 hour opioid (fentanyl) use. This study is conducted in Tuen Mun hospital (TMH) and Pok Oi hospital (POH) in Hong Kong. Patient are recruited for the study during pre-anaesthetic assessment, and they are counselled for risk of general anaesthesia and erector spinae plane block (i.e. local infection/bleeding, injury to neighbouring structure, local anaesthetic toxicity).

DETAILED DESCRIPTION:
After a pilot study regarding opioid use for patient after THR, the sample size for either treatment or control arm is calculated to be 35 patients per group to achieve adequate power to detect such a difference.

Sealed opaque envelopes with allocation inside is prepared forehand and is subsequently drawn on the day of surgery. The attending anaesthetist receives the envelope right before induction, and opens the envelope after the patient is put under general anaesthesia (GA). If the operation is cancelled or the patient cannot use PCA post-operatively (e.g. post-operative mechanical ventilation) or post-operative delirium), the envelope is put back into the pool.

After the patient is put under GA and turned lateral, the envelope is opened. For the treatment arm, lumbar ESP block is performed while for control arm no regional anaesthesia is performed nor saline is injected into the ESP. Before proceeding to ESP block, the back is cleaned with aseptic technique and draped. 40 mL of 0.25% levobupivacaine (or maximum of 2mg/kg body weight made up to same volume) is injected into the ESP.

After the injection, the surgeon is told not to infiltrate any local anaesthetics into the incision site or the wound. Intra-operatively, intravenous fentanyl is given as the only analgesic by the attending anaesthetist. Post-operatively, the patient is given fentanyl PCA of standard setting anaesthetist). The patient is also given all the pre-operative regular oral analgesic agents post-operatively, including paracetamol, NSAID, gabapentinoid and/or weak opioid (DF118 or tramadol).

The patient is assessed by an independent assessor from the acute pain service team 24 hours after the operation, who is blinded from the allocation result. Primary outcomes, that are post-operative 12 and 24 hour PCA fentanyl use and pain score in numeric rating scale (NRS) from 0 to 10 at rest and upon mobilisation are assessed and documented in the electronic system and also the patient chart. Secondary outcomes like presence/absence of PONV and knee flexion power in MRC scale are also noted.

The data are collected by the investigator and input to Excel 2003. 2-sided student's t test is used to compare the primary outcomes and also knee flexion power between treatment group and control group, while the rate of PONV between two groups is compared by Chi-square test. Multi-variate regression is done to control for the effect of oral analgesics on study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >=18)
* American Society of Anesthesiologists (ASA) class 1-3
* primary elective unilateral THR
* understand and accept the risk for general anaesthesia and ESP block
* counselled of post-operative patient controlled analgesia (PCA) and deemed fit for its use.

Exclusion Criteria:

* emergency THR
* bilateral THR
* revision THR
* THR done under neuraxial technique (e.g. spinal anaesthesia, combined spinal epidural anaesthesia)
* Patient with contraindication for ESP block (i.e. patient refusal, injection site infection or spine pathology/surgery, coagulopathy with international normalised ratio (INR) > 1.4 and thrombocytopenia < 75 x 10^9/L)
* patient who are mentally incompetent
* severe obesity (Body Mass Index >= 35)
* severe obstructive sleep apnea syndrome (Apnoea hypopnoea index >= 30, no matter on treatment or not)
* patient on regular strong opioid (e.g. morphine, oxycodone, methadone, buprenorphine, fentanyl)
* patient who have undergone hip neurolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony KT Ng, Study Director — Department of Anaesthesia and Intensive Care, Tuen Muen Hospital
Locations (1):
- Department of Anaesthesia and Intensive Care, Tuen Mun Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
data including patient number, age, gender, ASA class, anaesthetic technique, assignment, 24 hour fentanyl use, pain score, PONV and knee flexion power are available upon request by email to principal investigator
Supporting Information: Study Protocol
Time Frame: data available up to 1 year after completion of study
Access Criteria: for validation of study results or for compilation of systemic review/meta-analysis

REFERENCES:
- [Background] Switon A, Wodka-Natkaniec E, Niedzwiedzki L, Gazdzik T, Niedzwiedzki T. Activity and Quality of Life after Total Hip Arthroplasty. Ortop Traumatol Rehabil. 2017 Oct 31;19(5):441-450. doi: 10.5604/01.3001.0010.5823. PMID 29154234
- [Background] Chandrasekaran S, Ariaretnam SK, Tsung J, Dickison D. Early mobilization after total knee replacement reduces the incidence of deep venous thrombosis. ANZ J Surg. 2009 Jul;79(7-8):526-9. doi: 10.1111/j.1445-2197.2009.04982.x. PMID 19694660
- [Background] Zhang XY, Ma JB. The efficacy of fascia iliaca compartment block for pain control after total hip arthroplasty: a meta-analysis. J Orthop Surg Res. 2019 Jan 25;14(1):33. doi: 10.1186/s13018-018-1053-1. PMID 30683117
- [Background] Tulgar S, Ermis MN, Ozer Z. Combination of lumbar erector spinae plane block and transmuscular quadratus lumborum block for surgical anaesthesia in hemiarthroplasty for femoral neck fracture. Indian J Anaesth. 2018 Oct;62(10):802-805. doi: 10.4103/ija.IJA_230_18. PMID 30443064
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Gasanova I, Alexander JC, Estrera K, Wells J, Sunna M, Minhajuddin A, Joshi GP. Ultrasound-guided suprainguinal fascia iliaca compartment block versus periarticular infiltration for pain management after total hip arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2019 Feb;44(2):206-211. doi: 10.1136/rapm-2018-000016. PMID 30700615
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] World Health Organization. ICD-11: International Classification of Diseases (11th Revision). 2019
- [Background] Australian and New Zealand College of Anaesthetists. PM01 (Appendix 2): Opioid dose Equivalence - Calculation of Oral Morphine Equivalent Daily Dose (oMEDD). 2021.
- [Background] Austin PC. Balance diagnostics for comparing the distribution of baseline covariates between treatment groups in propensity-score matched samples. Stat Med. 2009 Nov 10;28(25):3083-107. doi: 10.1002/sim.3697. PMID 19757444
- [Background] Chow SC, Shao J, Wang H. Sample Size Calculations in Clinical Research. 2nd ed. Chapman & Hall/CRC; 2008.
- [Background] Iwanaga J, Simonds E, Schumacher M, Yilmaz E, Altafulla J, Tubbs RS. Anatomic Study of the Superior Cluneal Nerve and Its Related Groove on the Iliac Crest. World Neurosurg. 2019 May;125:e925-e928. doi: 10.1016/j.wneu.2019.01.210. Epub 2019 Feb 11. PMID 30763748
- [Background] Davies A, Crossley A, Harper M, O'Loughlin E. Lateral cutaneous femoral nerve blockade-limited skin incision coverage in hip arthroplasty. Anaesth Intensive Care. 2014 Sep;42(5):625-30. doi: 10.1177/0310057X1404200513. PMID 25233177
- [Background] Tomlinson J, Ondruschka B, Prietzel T, Zwirner J, Hammer N. A systematic review and meta-analysis of the hip capsule innervation and its clinical implications. Sci Rep. 2021 Mar 5;11(1):5299. doi: 10.1038/s41598-021-84345-z. PMID 33674621
- [Background] Gadsden J, Warlick A. Regional anesthesia for the trauma patient: improving patient outcomes. Local Reg Anesth. 2015 Aug 12;8:45-55. doi: 10.2147/LRA.S55322. eCollection 2015. PMID 26316813
- [Background] Oh SK, Lim BG, Won YJ, Lee DK, Kim SS. Analgesic efficacy of erector spinae plane block in lumbar spine surgery: A systematic review and meta-analysis. J Clin Anesth. 2022 Jun;78:110647. doi: 10.1016/j.jclinane.2022.110647. Epub 2022 Jan 11. PMID 35030493
- [Background] Kokar S, Ertas A, Mercan O, Yildirim FG, Tastan OA, Akgun K. The lumbar erector spinae plane block: a cadaveric study. Turk J Med Sci. 2022 Feb;52(1):229-236. doi: 10.3906/sag-2107-83. Epub 2022 Feb 22. PMID 34773689
- [Background] Soffin EM, Okano I, Oezel L, Arzani A, Sama AA, Cammisa FP, Girardi FP, Hughes AP. Impact of ultrasound-guided erector spinae plane block on outcomes after lumbar spinal fusion: a retrospective propensity score matched study of 242 patients. Reg Anesth Pain Med. 2022 Feb;47(2):79-86. doi: 10.1136/rapm-2021-103199. Epub 2021 Nov 17. PMID 34795027
- [Background] Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, Hollmann MW, Poepping DM, Schnabel A, Kranke P. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009642. doi: 10.1002/14651858.CD009642.pub3. PMID 29864216
- [Background] Abdelnasser A, Zoheir H, Rady A, Ramzy M, Abdelhamid BM. Effectiveness of ultrasound-guided erector spinae plane block for postoperative pain control in hip replacement surgeries; A pilot study. J Clin Anesth. 2020 Jun;62:109732. doi: 10.1016/j.jclinane.2020.109732. Epub 2020 Jan 25. No abstract available. PMID 31986435
- [Derived] Chan A, Ng TKT, Tang BYH. Single-Shot Lumbar Erector Spinae Plane Block in Total Hip Replacement: A Randomized Clinical Trial. Anesth Analg. 2022 Oct 1;135(4):829-836. doi: 10.1213/ANE.0000000000006162. Epub 2022 Aug 1. PMID 35913722

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 36 | 35
Completed | 35 | 35
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.5) | 64.7 (10.2) | 64.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 35 | 70
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Score in Numeric Rating Scale (NRS) From 0 (no Pain) to 10 (Extreme Pain)
Description: at rest
Time Frame: First post-operative day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
score on a scale | 3 [0 to 5] | 3 [0 to 4.5]

2. Primary Outcome: Post-operative Pain Score in Numeric Rating Scale (NRS) From 0 (no Pain) to 10 (Extreme Pain)
Description: upon mobilisation
Time Frame: First post-operative day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
score on a scale | 7 [6 to 8] | 7 [4.5 to 8.5]

3. Primary Outcome: Post-operative 12 Hour Fentanyl (Intravenous Patient-controlled Analgesia) Use
Description: in microgram
Time Frame: 12 hour post-operatively
Measure: Median (Inter-Quartile Range); unit: Microgram
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
Microgram | 210 [140.5 to 363] | 165 [77.5 to 330.5]

4. Primary Outcome: Post-operative 24 Hour Fentanyl (Intravenous Patient-controlled Analgesia) Use
Description: in microgram
Time Frame: 24 hour post-operatively
Measure: Median (Inter-Quartile Range); unit: Microgram
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
Microgram | 409 [221 to 636.5] | 349 [114 to 626.5]

5. Secondary Outcome: Post-operative Nausea and Vomiting (PONV)
Description: either presence of nausea or vomiting of any degree counted as yes
Time Frame: First post-operative day
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
Participants | 11 | 10

6. Secondary Outcome: Knee Flexion Power (Operative Side)
Description: measured in medical research council (MRC) grade with 0 being no movement to maximum of 5 meaning normal power
Time Frame: First post-operative day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
score on a scale | 3 [2 to 4] | 3 [2 to 3]

ADVERSE EVENTS:
Time Frame: 24 hour post-operatively
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 1/35 | 0/35
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=35) | Control (N=35)
Prolonged motor block (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Prolonged lower limb weakness which resolved spontaneously after 3 weeks

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT04388553/Prot_SAP_001.pdf